CLINICAL TRIAL: NCT01545869
Title: Efficacy and Safety of Fractional Carbon Dioxide Laser for Treatment of Facial Freckles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Pr. Bakr Mohamed Elzawahry, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fractional CO2 in freckles
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Freckles
Keywords: carbon dioxide laser; fractional resurfacing; freckles; melanosis
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fractional carbon dioxide laser (Experimental)
  Interventions: Procedure: Fractional carbon dioxide laser

INTERVENTIONS:
Procedure: Fractional carbon dioxide laser — SmartXide fractional carbon dioxide laser (DEKA, Florence, Italy). Parameters adjusted for: Power 20 watts, spacing 200 µsec, dwell time 300 µm, stacks 1.
  Other Names: Ablative fractional laser resurfacing

SUMMARY:
Freckles are clusters of melanin in the superficial epidermis. They affect mostly face and sun exposed areas, and appear as flat brown or red macules that fade in winter, usually in a fair complexion patient, but may be present in other skin types.

The gold standard in the industry for non-surgical facial rejuvenation, removal of wrinkles, pigmentation, and general sun damage has been the carbon dioxide (CO2) laser since the mid 1990s. The traditional CO2 laser was very effective, however it fell out of favor because it required general anesthesia. It also had a prolonged recovery time. Over the last several years, advances in technology known as fractional resurfacing has made the CO2 laser popular again: Fractional CO2 laser treatment is one of the newest laser rejuvenation technology. It proved successful in treatment of melasma, one of the pigmented dermatoses. To the best of our knowledge, based on a thorough search of literature, no clinical studies assessing fractional CO2 laser in treatment of freckles could be retrieved.

ELIGIBILITY:
Inclusion Criteria:

* -Patients affected with facial freckles.
* Age: 10 years or more

Exclusion Criteria:

* Patients younger than 10 years old.
* Patients aged 10-21 years who can not provide a written consent of parents or legal guardian.
* Patients with known tendency to keloid or hypertrophic scar formation.
* Patients receiving treatment with systemic retinoids or having stopped their course since less than six months duration.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
treatment success | One month
  reduction of freckles number and color density more than 50% in comparison to pre-treatment digital photos

SECONDARY OUTCOMES:
Treatment safety | three months
  Absence of irreversible changes in color and texture of the facial skin, that can cause patient dissatisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Bakr M Elzawahry, MD, Study Chair — Cairo University; Vanessa G Hafez, MD, Principal Investigator — Cairo University; Aya Fahim, MBBCh, Principal Investigator — Cairo University
Locations (1):
- Dermatology department - faculty of medicine- Cairo University, Cairo, Egypt